CLINICAL TRIAL: NCT00552461
Title: Prospective Open-Label Trial of Rituximab for Primary Pulmonary Alveolar Proteinosis
Brief Title: Prospective Trial of Rituximab for Primary Pulmonary Alveolar Proteinosis
Acronym: PAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Malur, Anagha, Research Director, Division of Pulmonary, Critical Care and Sleep Medicine, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U2990s
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Alveolar Proteinosis; Primary Disease
Keywords: Pulmonary alveolar proteinosis; Primary Pulmonary alveolar proteinosis; Rituximab; Idiopathic; Symptomatic; GM-CSF Antibody
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — IV, 1000 mg, two weeks, 2 times
  Other Names: Rituxan; MabThera

SUMMARY:
The purpose of this study is to determine whether the use of rituximab is effective in treating pulmonary alveolar proteinosis by leading to an improvement in lung function and disease status.

DETAILED DESCRIPTION:
The goal of this study is to conduct a prospective, open-label 6-month trial of rituximab in patients who present with symptomatic primary or idiopathic PAP. A total of 10 subjects with primary PAP will be enrolled over 12 months at East Carolina University. Patients over age 18 with a clinical diagnosis of moderate symptomatic idiopathic PAP, established by appropriate clinical history, radiographic and physiologic findings, presence of circulating anti-GM-CSF antibody, and confirmatory findings on bronchoscopy with bronchoalveolar lavage and/or open-lung biopsy will be recruited. Patients with newly diagnosed PAP or established disease may be considered for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary PAP (new or chronic) with presence of anti-GM-CSF antibody
* Moderately symptomatic disease with PaO2 <70 on room air and on less than 6 L/min oxygen
* Able to give written informed consent and comply with the requirements of the study
* Adequate renal and liver function
* Negative serum pregnancy test (for women of child bearing age) and on acceptable birth control during and after study completion

Exclusion Criteria:

* Severe PAP and requires in-patient care and more urgent therapy with bilateral whole lung lavage
* Treatment with any investigational agent within 4 weeks of screening
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of HIV, recurrent significant infection or recurrent bacterial infections
* Known active bacterial, viral, fungal, mycobacterial, or other infection
* Ongoing use of high dose steroids (>10mg/day) or unstable steroid dose
* Significant cardiac or pulmonary disease or blood disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluate symptomatic, physiologic and radiographic effects of therapy | 6-months

SECONDARY OUTCOMES:
Evaluate the overall tolerability of therapy and the requirement for therapeutic whole-lung lavage | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Mani S Kavuru, MD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

REFERENCES:
- [Derived] Kavuru MS, Malur A, Marshall I, Barna BP, Meziane M, Huizar I, Dalrymple H, Karnekar R, Thomassen MJ. An open-label trial of rituximab therapy in pulmonary alveolar proteinosis. Eur Respir J. 2011 Dec;38(6):1361-7. doi: 10.1183/09031936.00197710. Epub 2011 Apr 8. PMID 21478218
- See also: East Carolina University Division of Pulmonary — http://www.ecu.edu